CLINICAL TRIAL: NCT06510829
Title: Comparative Study Between Effect of Bleomycin Intralesional Injection And Application of Diode Laser on Infantile Hemangioma.
Brief Title: Comparison Between Diode Laser and Bleomycin in Treatment of Hemangioma
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kerolos Fayez, Kerolos Fayez Youakeem, Assiut University
Other Study IDs: Diode laser hemangioma
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Bleomycin Adverse Reaction
MeSH Terms: interventions — Lasers, Semiconductor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Group will be treated with intralesional bleomycin injection
- Group b: Group will be treated with application of diode laser
  Interventions: Device: Diode laser

INTERVENTIONS:
Device: Diode laser — Application of laser waves on the lesion
  Groups: Group b

SUMMARY:
Assessment of the Effectiveness of Bleomycin Intralesional Injection and Diode Laser on Management of Infantile Hemangioma., with regard to :

* Clinically based on Change in the Size and Color of Hemangioma.
* Ultrasonography considering Vascularity ,Echogenicity , Height , and Morphology .
* Comparison of Complications associated with Bleomycin and Diode Laser.

ELIGIBILITY:
Inclusion Criteria:

* Age between 3 Months and 1 Year old.
* Non Complicated Infantile Hemangioma

Exclusion Criteria:

* Younger than 3 Months or older than 1 Year.
* Complicated Infantile Hemangioma

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Comparative Study Between Effect of Bleomycin Intralesional Injection And Application of Diode Laser on Infantile Hemangioma .
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Effect of diode laser on hemangioma | 3 years

IPD SHARING:
Plan to Share IPD: Undecided